CLINICAL TRIAL: NCT07011498
Title: Connecting Through Choir Singing: Dementia Choirs to Reduce Loneliness in Home-dwelling Persons Living With Dementia and Their Caregivers - a Crossover Study
Brief Title: Dementia Choirs for Social and Psychological Wellbeing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Academy of Music (Other)
Collaborators: Oslo Municipality (Other Government); Institute of Clinical Medicine, University of Oslo (Unknown); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 828898
Record Dates: First submitted 2025-03-10; First posted 2025-06-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Informal Caregivers (Family and Friends)
Keywords: Dementia; Choir; Loneliness; Music therapy
MeSH Terms: conditions — Dementia | interventions — Singing; Music Therapy

STUDY DESIGN:
Intervention Model Description: The study has a single group model in a crossover design. In the study, participants will be recruited to participate in dementia choirs. The choirs will be divided into two groups. Participants in each group will complete all assessments at the same timepoints but receive choir activity at different times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia choir (Experimental)
  Interventions: Other: Dementia choir

INTERVENTIONS:
Other: Dementia choir — Music therapy informed dementia choirs will be delivered once a week. Rehearsals last app. 2 hours, including a social break. Each choir will be led by 1 conductor and 1 accompanist. The choir leaders will have relevant professional qualifications that supplement each other, such as a music therapist, music pedagogue, conductor, singer, singing teacher, or health care professional with additional music competence. They will be trained by the research team to deliver the choirs in a dementia friendly and music therapy informed way. In addition, the choir leaders will receive supervision from the research team throughout the intervention periods. The choirs will involve volunteers to assist during rehearsals and breaks. The volunteers will also receive training on how to support the choir participants in a dementia friendly way.
  Other Names: choir; singing; music therapy

SUMMARY:
Loneliness is common in both persons living with dementia and their informal caregivers, and a factor negatively affecting disease progression, health and wellbeing. However, intervention studies to address loneliness show inconsistent effects. This study aims to evaluate effect of a community-based group intervention - music therapy informed dementia choirs - on loneliness for home-dwelling people with dementia and their informal caregivers. We will recruit participants to five dementia choirs with 15-20 people in each and implement a crossover study with measures collected at four timepoints: baseline, 12-week follow up, 22-week follow-up after an extended summer holiday, and 12-week follow-up after the summer holiday. The primary outcome, loneliness in participants living with dementia, will be measured using the De Jong Gierveld loneliness scale. Secondary outcomes will be depression, experience of meaning in life, apathy and mood for the participants living with dementia, and loneliness and caregiver burden for the informal caregivers. Cognition in the participants living with dementia, measured with the RUDAS assessment tool, will be included as a control variable. Further, measurements to evaluate the cost effectiveness of the choir intervention will be included, and qualitative data collected through semi-structured interviews to explore the experiences and possible impacts of the choir intervention in the participants' lives.

ELIGIBILITY:
Inclusion Criteria:

* Dementia diagnosis (Alzheimers, Lewy-body, fronto-temporal, vascular, mixed, Parkinson's dementia) or cognitive impairment as reported by the person themselves/their caregiver
* Informal caregiver of participant with dementia: A person who has a close relationship with a recruited choir participant living with dementia. A close relationship may for instance be a spouse/partner, sibling, adult child, friend, niece or nephew
* Living at home in the community

Exclusion Criteria:

* Significant hearing impairment that is not resolved through the use of a hearing aid device and limit their capacity to enjoy musical experiences.
* Formal (paid) caregiver of participant with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in degree of loneliness in participants with dementia at 12 weeks (primary), 22 weeks and 36 weeks follow up | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised questionnaire the De Jong Gierveld 6-item Loneliness Scale

SECONDARY OUTCOMES:
Change from baseline in degree of depression in participants with dementia to 12-week (primary timepoint), 22-week and 26-week follow up | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised questionnaire Geriatric Depression Scale Short-Version, GDS-15.
Change from baseline in degree of self-reported meaning in life in participants with dementia to 12-week (primary timepoint), 22-week and 26-week follow up | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised questionnaire The Meaning in Life Questionnaire Short Form (MLQ-SF)
Change from baseline in degree of apathy in participants with dementia to 12-week (primary timepoint), 22-week and 26-week follow up | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised questionnaire Apathy Evaluation Scale - Informant Version, reported by informal caregivers as proxy.
Change from baseline in degree of loneliness in informal caregivers of participants with dementia to 12-week (primary timepoint), 22-week and 26-week follow up | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised questionnaire The De Jong Gierveld 6-item Loneliness Scale measuring degree of self-reported loneliness.
Change from baseline in degree of caregiver burden to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up. | From baseline to 12-week follow up (primary timepoint), 22-week follow up and 36-week follow up.
  Measured by the standardised self-reported questionnaire Relative's Stress Scale (RSS)
Change of mood in participant with dementia from before to after choir rehearsals | From before to after rehearsals for rehearsals 2, 6 and 11 (per choir).
  Measured by tha standardised questionnaire The Dementia Mood Picture Test completed immediately before and after selected choir rehearsals (rehearsal 2, 6 and 11).

OTHER OUTCOMES:
Change from baseline in cognition of participants with dementia to 12-week and 36-week follow up | Entire intervention period comprising three measurements (baseline, 12-week follow-up, and final 12-week follow-up after an extended summer holiday)
  The Rowland Universal Dementia Assessment Scale (RUDAS), A Multicultural Cognitive Assessment Scale is included as a control variable.
Caregiver experience of choirs as a relief or a burden | At 36-week follow-up and during prolonged intervention after quantitative assessments
  Collected through a short 5-point Likert scale questionnaire asking them whether they experience the choir as a relief or a burden.
Change from baseline in Quality of life in participants with dementia, Quality-adjusted life-years to 12-week follow up | From baseline to 12-week follow up
  Measured by the EuroQol instrument (EQ-5D-5L) completed by informal caregiver as proxy.
Resource use in dementia care | From baseline to end of the first 12 week intervention period.
  The standardised instrument Resource utilisation in dementia (RUD) will be used to collect data about formal and informal care. The RUD assesses resource use about both the person living with dementia and the caregiver, including time expended in different daily tasks.
Rehearsing at home | Entire intervention from second measurement (12-week follow-up, 22-week follow-up after an extended summer holiday (lasting 8 weeks), and 12-week follow-up after the summer holiday)
  A self-completed questionnaire about whether they rehearse at home, and if so, how often
Participants experiences of choir singing | Qualitative interviews will be conducted between 36-week follow-up and study completion.
  Qualitative interviews with a selection of participants about their experiences of singing in the choir.
Adherence to intervention | Entire intervention period comprising four measurements (baseline, 12-week follow-up, 22-week follow-up after an extended summer holiday (lasting 8 weeks), and 12-week follow-up after the summer holiday)
  Participants' adherence by registering their attendence at choir rehearsals.
Adverse events | From baseline through study completion, app. 1 year
  Information about adverse events will collected throughout the intervention periods. Participants will be asked about any adverse events they may have experienced, including hospitalisations, unexpected health care appointments or negative responses to the intervention.
Change from baseline in Quality of life in informal caregivers of participants with dementia, Quality-adjusted life-years to 12-week follow up | From baseline to 12-week follow up
  Measured by the EuroQol instrument (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Kjersti Johansson, PhD, Principal Investigator — Norwegian Academy of Music
Locations (1):
- Norwegian Academy of Music, Oslo, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No